CLINICAL TRIAL: NCT05372510
Title: A Pilot Study to Evaluate the Feasibility of Identifying, Enrolling and Following Acute and Early HIV-1 Infected Individuals.
Brief Title: Feasibility of Identifying, Enrolling and Following Acute and Early HIV-1 Infected Individuals.
Acronym: KILGORIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MRC/UVRI and LSHTM Uganda Research Unit (Other)
Collaborators: International AIDS Vaccine Initiative (Network)
Responsible Party: Principal Investigator, Dr. Andrew Obuku, SCIENTIST, MRC/UVRI and LSHTM Uganda Research Unit
Other Study IDs: RGAO190401
Record Dates: First submitted 2022-05-05; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Acute Human Immunodeficiency Virus Type I Infection
Keywords: HIV-1, immune responses, cell death, acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — PBMCs will be stored. plasma, serum, paxgene tubes will be stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is only between peak viremia and viral setpoint in natural acute HIV-1 infection that the immune response overwhelms viral replication resulting in a plasma viral load decline. The aim will be to characterize these immune responses, how they develop and their progeny. This will require the need to identify HIV-1 infected individuals before peak viremia and follow them to post viral setpoint.

This protocol describes a pilot study to evaluate the feasibility of identifying, enrolling and following acute and early HIV-1 infected individuals from voluntary counselling and testing centres in Masaka, Bukomansimbi, Kalungu, Lwengo, Sembababule and Lyantonde districts.

ELIGIBILITY:
Inclusion Criteria:

* Females and males.
* Able and willing to provide informed consent.
* Willing to undergo HIV testing using GeneX pert Viral Load assay.
* Able and willing to provide accurate locator information for tracking purposes and willing to be contacted by study staff.
* Willing to complete interviewer administered questionnaires on risk factors and if infected, questions related to the route and timing of exposure.

Exclusion Criteria:

Has any condition that in the opinion of the principal investigator or designee, would preclude provision of informed consent, or otherwise interfere with achieving the study objectives.

* Participation in a current clinical trial unless approved by the investigators and IAVI medical monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any females and males between 18years - No limit.
  * Able and willing to provide informed consent.
  * Willing to undergo HIV testing using GeneX pert Viral Load assay.
  * Able and willing to provide accurate locator information for tracking purposes and willing to be contacted by study staff.
  * Willing to complete interviewer administered questionnaires on risk factors and if infected, questions related to the route and timing of exposure.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
To measure the number of individuals who are Genexpert HIV Viral load assay positive and Alere Determine HIV-1/2 Negative. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: ANDREW OBUKU, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- MRC/UVRI & LSHTM, Uganda Research Unit,Masaka station, Masaka, Uganda